CLINICAL TRIAL: NCT00845325
Title: Early Motion Following Carpal Tunnel Release, a Randomized Control Trial
Brief Title: Early Motion Following Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Stephen Colbert, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1108957
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel release; Rehabilitation; Early motion
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — One-Carbon Group Transferases; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group One (Active Comparator): The first group (early motion) will have a bulky dressing placed at the time of surgery. They will be instructed to remove the dressing on the first postoperative day and to place a band-aid over the incision. A set of non-weight bearing "stretching" exercises will be explained on the day of surgery and instructions with diagrams sent home with the patient. They will begin these exercises on the day after surgery and perform them three times daily for two weeks. The patients will have no restrictions concerning activity or return to work.
  Interventions: Behavioral: Group One
- Behavorial Control Group Two (Other): The second group will have wrist immobilization splints placed at the time surgery. The thumb and fingers will not have limited motion in this splint. Due to the splint placement, the patients will be restricted from using that hand during its implementation. One week following surgery the splint will be removed and the patient will be instructed to begin activity without restriction.
  Interventions: Behavioral: Control Group Two

INTERVENTIONS:
Behavioral: Group One — They will begin exercises on the day after surgery and perform them three times daily for two weeks. The patients will have no restrictions concerning activity or return to work.
  Other Names: early motion/rehabilitation
  Arms: Group One
Behavioral: Control Group Two — The patients will be restricted from using that hand during its implementation. One week following surgery the splint will be removed and the patient will be instructed to begin activity without restriction.
  Other Names: Delayed rehabilitation
  Arms: Behavorial Control Group Two

SUMMARY:
To objectively and subjectively assess two modes of commonly employed rehabilitation and confirm a superior method to treat patients following carpal tunnel release.

One of the problems following carpal tunnel release (CTR) for carpal tunnel syndrome, and all hand surgeries, is the debilitation in the postoperative period. This relates to muscle atrophy and joint stiffness due to immobilization or relative inactivity in the postoperative period. Specifically, patients suffer increased days off from work, lost wages, and difficulties with activities of daily living affecting the patient and society at large. CTR is a very common procedure in hand surgery making it easy to study and important to optimize the postoperative care.

DETAILED DESCRIPTION:
The surgical procedure, carpal tunnel release, will be performed in a standard open fashion. In a random fashion, the patients will be placed into either of two rehabilitation groups following CTR with specifically different postoperative instructions after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of carpal tunnel syndrome
* Recommended for carpal tunnel release

Exclusion Criteria:

* Severe thenar weakness
* proximal neuropathy of the same arm.
* generalized peripheral neuropathy
* active psychiatric disorder
* chronic renal failure require dialysis
* reflex sympathetic dystrophy
* previous injury of affected wrist or median nerve
* simultaneous ipsilateral upper extremity surgery
* carpal tunnel syndrome with acute injury

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
days to return to activities of daily living, return to work, grip strength, pinch strength, digital sensibility, subjective pain control, number of pain pills used, grading of success,and any complications encountered. | 1 week, 3 weeks, 3 months, and 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H Colbert, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No